CLINICAL TRIAL: NCT07381946
Title: Clinical Study on Bilateral High-frequency Repetitive Transcranial Magnetic Stimulation Combined With Swallowing Training for Patients With Dysphagia After Extubation
Brief Title: High-frequency Repetitive Transcranial Magnetic Stimulation for Patients With Dysphagia After Extubation
Acronym: Dysphagia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wuhan University (Other)
Responsible Party: Principal Investigator, Qing Shu, associate chief physician, Wuhan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025169K
Record Dates: First submitted 2026-01-09; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Post-extubation Dysphagia
Keywords: Dysphagia; Extubation failure; repetitive transcranial magnetic stimulation
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding After the intervention allocation, the participants and data analysts will be blinded. This is a single - blinded, randomized, parallel - controlled study focusing on rTMS. In the rTMS group, a 20 - minute magnetic stimulation will be applied to the target brain area.. Before the final code - breaking, data analysts won't know the group to which the data they are analyzing belongs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- a bilateral high-frequency repetitive transcranial magnetic stimulation plus swallowing training (Experimental)
  Interventions: Behavioral: Swallowing training; Device: a bilateral high-frequency repetitive transcranial magnetic stimulation
- Swallowing training plus No intervention (Placebo Comparator)
  Interventions: Behavioral: Swallowing training; Other: No intervention

INTERVENTIONS:
Behavioral: Swallowing training — Swallowing training includes facial function training, sensory stimulation training, and airway protection techniques.
Device: a bilateral high-frequency repetitive transcranial magnetic stimulation — The interventional targets were the key cortical brain regions identified in preliminary studies, with stimulation applied to the bilateral oral and tongue regions.Parameters included a figure-of-8 coil, 10 Hz frequency, 5-second stimulation duration,55-second inter-train intervals, 10 repetitions, totaling 500 pulses per session, with each session lasting 10 minutes. Swallowing Training commenced within 10 minutes post-rTMS, following the same duration and intensity as the Swallowing Training Group . The treatment was conducted three days.
  Arms: a bilateral high-frequency repetitive transcranial magnetic stimulation plus swallowing training
Other: No intervention — No intervention methods
  Arms: Swallowing training plus No intervention

SUMMARY:
Post-extubation dysphagia (PED) is characterized by a range of clinical manifestations, including absence of visible swallowing effort, coughing or choking following liquid intake, and post-swallowing dysarthria. These impairments may lead to severe complications such as aspiration pneumonia, electrolyte disturbances, and malnutrition. Currently, the majority of hospitals both domestically and internationally have not implemented routine screening for PED or standardized swallowing rehabilitation programs, and research on the recovery of swallowing function in PED remains limited. This study aims to investigate the therapeutic efficacy of bilateral high-frequency repetitive transcranial magnetic stimulation (rTMS) combined with conventional swallowing training in patients with PED, and to evaluate the influence of oral feeding on functional recovery and the incidence of pneumonia.

The study design is a single-center, randomized, single-blind, parallel-controlled trial. Participants with PED will be randomly assigned to either a swallowing training group or a bilateral high-frequency repetitive transcranial magnetic stimulation plus swallowing training group.The primary outcome measure is the Functional Oral Intake Scale (FOIS) score，which assesses oral feeding ability.Secondary outcomes include the Wakada Drinking Water Test(WST),degree of swallowing difficulty(GUSS),the incidence rate of pneumonia and length of stay.These secondary outcomes will provide a comprehensive evaluation of swallowing ability and hospitalization effects.

Random grouping was conducted within 4 hours after extubation, and the treatment began within 2 hours and lasted for 3 consecutive days.Each rTMS session will target key brain regions.Swallowing training includes facial function training, sensory stimulation training, and airway protection techniques.The observation group received bilateral high-frequency transcranial magnetic stimulation in addition to the swallowing training.The data will be collected before and after the treatment.The primary outcome, FOIS score, will be used to assess the overall improvement in oral feeding ability.WST and GUSS data will be collected to evaluate a comprehensive evaluation of swallowing ability.The incidence rate of pneumonia and length of stay will be used to assess change in side effects.

Statistical analyses will be performed using SPSS 22.0. Data will be presented as mean ± standard deviation. Between-group differences will be compared using independent samples t-tests.

The study timeline spans from September 2025 to December 2026, including participant recruitment, intervention implementation, data collection, and analysis, as well as manuscript drafting. This study aims to provide new insights into the treatment methods for PED and explore a new rehabilitation approach that can be used in the ICU, with the expectation of improving swallowing disorders and reducing complications.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years;
2. Tracheal intubation for more than 48 hours;
3. Clear consciousness at the time of assessment, able to understand and follow the simple instructions of the researchers;
4. Patients have dysphagia, and the Functional Oral Intake Scale (FOIS) assessment is at levels

Exclusion Criteria:

1. Previous history of dysphagia;
2. Undergoing tracheotomy;
3. History of epilepsy;
4. Having metal implants in the brain;
5. Implanted with a cardiac pacemaker;
6. Under absolute isolation (such as open or infectious pulmonary tuberculosis);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Functional Oral Intake Scale ，FOIS | Baseline (before treatment), 3 days after treatment
  The oral feeding ability was conducted using the Functional Oral Intake Scale (FOIS), which is divided into 7 levels. The higher the level, the better the oral intake ability.

SECONDARY OUTCOMES:
Wakada Drinking Water Test，WST | Baseline (before treatment), 3 days after treatment
  The swallowing function was evaluated using the WST. The classification ranges from level 1 to level 5. The higher the level, the poorer the drinking ability
degree of swallowing difficulty，GUSS | Baseline (before treatment), 3 days after treatment
  The GUSS is a widely used assessment tool for evaluating functional outcomes in dysphagia. It includes domains such as attention, spontaneous coughing, swallowing saliva, drooling, and voice.The direct swallowing test section involves screening for the swallowing of thickened food, liquid food, and solid food, respectively, to assess the situations of delayed swallowing, spontaneous coughing, drooling, and voice changes.The total score is 20 points, with 0 to 9 points indicating severe dysphagia; 10 to 14 points indicating moderate dysphagia; 15 to 19 points indicating mild dysphagia; and 20 points indicating no dysphagia.
length of stay | at discharge
  The earlier a patient is discharged, the less financial burden it will impose on them

OTHER OUTCOMES:
the incidence rate of pneumonia | 30 days after extubation
  A lower incidence of pneumonia indicates fewer complications

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan hospital of Wuhan University, Wuhan, Hubei 430070, Wuhan, Hubei, China

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-02): https://cdn.clinicaltrials.gov/large-docs/46/NCT07381946/Prot_SAP_000.pdf